CLINICAL TRIAL: NCT01734538
Title: Effects of 12 Weeks of Omega-3 Fatty Acid Supplementation on Metabolic and Physical Health Parameters in Older Adults
Brief Title: Effect of 12 wk of Omega-3 FA Supplementation on Metabolic and Physical Health Parameters in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Lawrence Spriet, Dr. Lawrence Spriet, University of Guelph
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 12OC014
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Effect of Omega-3 Fatty Acid Supplementation Physical Fitness

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Omega-3 Complete (Experimental): Oral ingestion of 3000 mg (5 capsules) of Omega-3 Complete (Jamieson Laboratories, Ltd., Windsor, Ontario, Canada) per day for 12 weeks.
  Interventions: Dietary Supplement: Omega-3 Complete
- Placebo Capsule (Placebo Comparator): Oral ingestion of 5 capsules of a placebo oil pill (Jamieson Laboratories Ltd., Windsor, Ontario, Canada) per day for 12 weeks
  Interventions: Dietary Supplement: Placebo capsule

INTERVENTIONS:
Dietary Supplement: Omega-3 Complete
  Arms: Omega-3 Complete
Dietary Supplement: Placebo capsule
  Arms: Placebo Capsule

SUMMARY:
The biological membranes that surround a cell and its organelles are important to the overall function of the cell. Fatty acids are the main structural components of a membrane, and the presence of certain fatty acids can alter a membrane's characteristics, which subsequently alters its function. Two fatty acids that are of particular interest to researchers are eicosapentanoic acid (EPA) and docosahexanoic acid (DHA). These omega-3 fatty acids have unique unsaturated structures, and their incorporation into biological membranes appears to elicit potent physiological effects. The body is unable to intrinsically synthesize these important fatty acids, so they must be obtained from the diet or through supplementation.

EPA and DHA supplementation has been reported to provide numerous positive health benefits, including decreased blood pressure and an improved blood lipid profile. Recent research in our laboratory has demonstrated in young men that resting metabolic rate was increased following a 12 week period of omega fatty acid supplementation of 3 g/day. Fat utilization was also increased and carbohydrate use was decreased both at rest and during a 1 hr moderate exercise challenge. These findings have positive implications for people who are interested in losing weight, but it not known whether these effects occur in older adults. With age, body composition changes (increase in fat mass and decrease in lean mass) occur which may negatively affect general health, particularly normal physical functioning and quality of living of the older adult. The potential role of omega 3 fatty acids to increase fat oxidation and increase resting metabolic rate may be a therapy for decreasing fat mass in the older adult. Research has suggested that omega 3 fatty acids may elicit an additional therapeutic role by reducing joint pain.

Another aspect of aging is a loss in lean body mass, which is associated with an attenuation of skeletal muscle protein synthesis in response to nutritional stimuli (amino acids and insulin). The weakened anabolic response is considered to be partly due to defects in the anabolic signaling cascade in the muscle. Research in older adults has reported an increase in muscle protein signaling with EPA and DHA supplementation in response to a nutritional challenge. However it is unknown whether the increase in protein signaling results in an eventual increase in lean body mass. The physical functioning of older adults is not only influenced by body composition changes, but also age-related neuronal changes that affect the velocity of axonal conduction and influence the ability of the muscle to generate torque and the rate at which the torque is developed. Muscular strength and functional capacity increases have been reported with chronic resistance exercise in a cohort of older women supplemented with EPA and DHA. However, the effect of EPA and DHA intake on physical strength in older adults with previously low EPA and DHA consumption, independent of exercise, is currently unknown.

Therefore, the purpose of this study is to determine the effects of 12 weeks of omega-3 supplementation at 3 g/day on metabolic and physical health parameters in community-dwelling older adults. We hypothesize that EPA and DHA supplementation will result in 1) a decrease in resting heart rate and blood pressure; 2) a more healthy blood profile; 3) an increase in resting metabolic rate; 4) a greater reliance on fat oxidation for energy both at rest and during exercise; and 5) a decrease in fat mass; and 6) an increase in lean mass, strength and physical function.

ELIGIBILITY:
Inclusion Criteria:

* 60 to 74 years of age
* Community-dwelling

Exclusion Criteria:

* Current or previous supplementation with omega-3's
* Average fish intake greater than one time per week
* Diagnosed heart condition
* Lightheadeness, shortness of breath, chest pain, numbness, fatigue, coughing, or wheezing during rest or at low to moderate physical activity
* Cardiovascular disease risk factors: family history of heart attacks, hypertension, hypercholesterolemia, diabetes mellitus, and smoking
* Allergies to lidocaine, fish/fish oil, gelatin, glycerin, or mixed tocopherols
* Currently taking any medications or supplements that may increase the chance of bleeding (e.g. Aspirin, Coumadin, Anti-inflammatories, Plavix, Vitamin C or E, high doses of garlic, gingko biloba, willow bark products)

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Change in resting heart rate from baseline | baseline and 12 weeks
Change in resting blood pressure from baseline | baseline to 12 weeks
Change in fasted blood triglyceride concentration from baseline | baseline to 12 weeks
Change in fasted blood cholesterol from baseline | baseline to 12 weeks
Change in blood c-reactive protein concentration from baseline | baseline to 12 weeks
Change in fasted blood low-density lipoprotein concentration from baseline | baseline to 12 weeks
change in fasted blood high-density lipoprotein concentration from baseline | baseline to 12 weeks
Change in fasted blood insulin concentration from baseline | baseline to 12 weeks
Change in fasted blood glucose concentration from baseline | baseline to 12 weeks
Change in whole body resting fat oxidation from baseline | baseline to 12 weeks
Change in whole body resting carbohydrate oxidation from baseline | baseline to 12 weeks
Change in whole body sub-maximal ecercise fat oxidation from baseline | baseline to 12 weeks
Change in whole body sub-maximal ecercise carbohydrate oxidation from baseline | baseline to 12 weeks
Change in resting metabolic rate from baseline | baseline to 12 weeks
Change in fat mass from baseline | baseline to 12 weeks
Change in lean mass from baseline | baseline to 12 weeks
Change in strength from baseline | baseline to 12 weeks
Change in physical function (balance) from baseline | baseline to 12 weeks

SECONDARY OUTCOMES:
Change in self-reported pain from baseline | baseline to 12 weeks
Change in self-reported overall health from baseline | baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence L. Spriet, PhD, Principal Investigator — The University of Guelph
Locations (1):
- The University of Guelph, Guelph, Ontario, Canada

REFERENCES:
- [Background] Kiecolt-Glaser JK, Belury MA, Andridge R, Malarkey WB, Hwang BS, Glaser R. Omega-3 supplementation lowers inflammation in healthy middle-aged and older adults: a randomized controlled trial. Brain Behav Immun. 2012 Aug;26(6):988-95. doi: 10.1016/j.bbi.2012.05.011. Epub 2012 May 26. PMID 22640930
- [Background] Rodacki CL, Rodacki AL, Pereira G, Naliwaiko K, Coelho I, Pequito D, Fernandes LC. Fish-oil supplementation enhances the effects of strength training in elderly women. Am J Clin Nutr. 2012 Feb;95(2):428-36. doi: 10.3945/ajcn.111.021915. Epub 2012 Jan 4. PMID 22218156
- [Background] Smith GI, Atherton P, Reeds DN, Mohammed BS, Rankin D, Rennie MJ, Mittendorfer B. Dietary omega-3 fatty acid supplementation increases the rate of muscle protein synthesis in older adults: a randomized controlled trial. Am J Clin Nutr. 2011 Feb;93(2):402-12. doi: 10.3945/ajcn.110.005611. Epub 2010 Dec 15. PMID 21159787
- [Background] Couet C, Delarue J, Ritz P, Antoine JM, Lamisse F. Effect of dietary fish oil on body fat mass and basal fat oxidation in healthy adults. Int J Obes Relat Metab Disord. 1997 Aug;21(8):637-43. doi: 10.1038/sj.ijo.0800451. PMID 15481762
- [Background] Delarue J, Labarthe F, Cohen R. Fish-oil supplementation reduces stimulation of plasma glucose fluxes during exercise in untrained males. Br J Nutr. 2003 Oct;90(4):777-86. doi: 10.1079/bjn2003964. PMID 13129446
- [Background] Peoples GE, McLennan PL, Howe PR, Groeller H. Fish oil reduces heart rate and oxygen consumption during exercise. J Cardiovasc Pharmacol. 2008 Dec;52(6):540-7. doi: 10.1097/FJC.0b013e3181911913. PMID 19034030
- [Background] Calder PC. n-3 Fatty acids and cardiovascular disease: evidence explained and mechanisms explored. Clin Sci (Lond). 2004 Jul;107(1):1-11. doi: 10.1042/CS20040119. PMID 15132735
- [Derived] Logan SL, Spriet LL. Omega-3 Fatty Acid Supplementation for 12 Weeks Increases Resting and Exercise Metabolic Rate in Healthy Community-Dwelling Older Females. PLoS One. 2015 Dec 17;10(12):e0144828. doi: 10.1371/journal.pone.0144828. eCollection 2015. PMID 26679702